CLINICAL TRIAL: NCT06913907
Title: Changes in Methotrexate Polyglutamate Concentrations When Changing From Oral to Subcutaneous Methotrexate Therapy in Methotrexate-naive Patients With Rheumatoid Arthritis: (COSMOS Study)
Brief Title: Changes in MTX-PG Concentrations During Subcutaneous MTX Therapy in Patients With Rheumatoid Arthritis(COSMOS Study)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Keio University (Other)
Collaborators: Eisai Co., Ltd. (Industry); Mebix Inc (Industry)
Responsible Party: Principal Investigator, Yuko Kaneko, professor, Keio University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N20240003
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MTX group (Other)
  Interventions: Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Methotrexate (MTX) — Single arm study

SUMMARY:
Methotrexate is known to exist intracellularly as methotrexate polyglutamate, which is formed by the addition of glutamic acid after absorption into the body.

The objective of this study is to measure the concentration of methotrexate polyglutamate in red blood cells and peripheral blood mononuclear cells after initiating methotrexate treatment in patients with rheumatoid arthritis who have no prior history of using methotrexate (either subcutaneous or oral formulations). Additionally, we aim to examine changes in methotrexate polyglutamate concentrations when switching from oral methotrexate to subcutaneous Metoject, as well as to investigate the relationship between methotrexate polyglutamate concentration and the efficacy and safety of the treatment. Another objective of this study is to evaluate whether switching to subcutaneous Metoject allows for an increased maximum tolerable dosage while maintaining safety.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients who were previously untreated with MTX, regardless of route of administration 2) Patients aged >=18 years at the time of informed consent 3) Patients who meet 2010 EULAR/ACR criteria 4) Patients who have disease activity of SDAI >11 at screening 5) Patients who were previously untreated with JAK inhibitor or bDMARDs 6) Female of child-bearing potential who can use appropriate contraceptive during the study and for at least one menstrual period after completion of MTX administration, female in whom time from menopause to informed consent is >=1 year, or female of no child-bearing potential through sterilization 7) Virile male who can use appropriate contraceptive during the study and for at least three months after completion of MTX administration 8) Patients who can adequately understand this study procedures, and voluntarily consent in writing to take part in this study

Exclusion Criteria:

* 1) Pregnant women or women who may be pregnant 2) Patients with a history of hypersensitivity to any ingredient of the study drug 3) Patients with serious hematologic and lymphatic disorders
* Patients with a history of myelodysplastic syndrome, aplastic anemia, or erythroblastoma
* Patients with a diagnosis or treatment of lymphoproliferative disease within the past 5 years
* Patients with significant leukopenia (white blood cell count <3000/mm3) or thrombocytopenia (platelet count <50000/mm3millimeter) 4) Patients with significant hepatic impairment
* Patients with acute or chronic active viral hepatitis B or C
* Patients diagnosed with cirrhosis
* Patients with other significant hepatic impairment (AST >150 U/L or ALT >150 U/L) 5) Patients with severe renal impairment The following criteria should be used as a reference.
* Dialysis patients or renal dysfunction correspon ding to renal glomerular filtration rate (GFR) <30 mL/min/1.73 m2 6) Patients who have pleural effusion or ascites 7) Patients who have active tuberculosis 8) Patients otherwise whom principal investigator/sub- investigator considered medically ineligible to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-10 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in MTX-PG concentrations in erythrocytes from baseline | From enrollment to the end of treatment at 24 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Keio University Hospital, Shinjuku-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No